CLINICAL TRIAL: NCT07110207
Title: Single-centre Descriptive Study of Taste in Frontotemporal Lobar Degeneration Through the Analysis of Taste Evoked Potentials
Acronym: FRONTAL-PEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JACQUIN 2025
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Frontotemporal Lobar Degeneration (FTLD)
MeSH Terms: conditions — Frontotemporal Lobar Degeneration | interventions — Hematologic Tests; Mental Status and Dementia Tests; Nutrition Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with frontotemporal lobar degeneration (Experimental)
  Interventions: Biological: Blood test; Other: Interrogation of the subject; Other: Cognitive assessment; Other: Nutritional assessment; Other: Taste tests; Other: Sucrose taste detection test

INTERVENTIONS:
Biological: Blood test — Metabolic measurements and measurements of hormones related to food intake
Other: Interrogation of the subject — Collection of socio-demographic data, medical and family history, medication
Other: Cognitive assessment — MMSE and MoCA cognitive tests
Other: Nutritional assessment — Anthropometric data (weight, height, BMI, waist circumference, hip circumference, android/gynoid ratio, triceps skinfold thickness, brachial circumference), bioelectrical impedance analysis (body fat percentage, lean body mass, body water percentage and bone mass in kg)
Other: Taste tests — Recording of PEGs in response to a sucrose solution (prepared beforehand)
Other: Sucrose taste detection test — Triangular test

SUMMARY:
The FRONTAL-PEG study focuses on taste perception in frontotemporal lobar degeneration (FTLD). This neurodegenerative disease, characterised by progressive loss of nerve cells, is the second leading cause of dementia after Alzheimer's disease.

Patients with FTLD often experience olfactory disorders (= sense of smell) and eating disorders: increased appetite, increased food intake and excessive consumption of sugary foods and snacking. This often leads to excessive weight gain. These eating disorders are still poorly understood at present.

In this context, we hypothesise that an alteration in the gustatory pathway - i.e. the way in which the brain perceives taste - could contribute to the eating disorders frequently observed in frontotemporal dementia (FTD), particularly in the marked attraction to sweet foods. We therefore wish to objectively evaluate the taste response to a sweet solution (sucrose) in patients with FTLD, using taste evoked potentials (TEPs). Taste evoked potentials are a reliable and reproducible technique for assessing brain activity in response to taste stimulation. One of their advantages is that they are non-invasive.

This study will document, for the first time in this disease, the characteristics of cortical (brain) processing of taste information.

The FRONTAL-PEG study is an interventional, regional, single-centre study conducted at the Dijon University Hospital, in collaboration with the CMRR (Memory, Resources and Research Centre) and the CSGA (Centre for Taste and Food Sciences).

All investigations are carried out at the CSGA (building adjacent to the Dijon University Hospital), with the exception of blood tests, which are carried out at the Dijon University Hospital.

The total duration of participation in the study is one morning. No follow-up is planned at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given their free and informed consent
* Person of legal age
* Fasting > 2 hours before PEG measurement
* Body Mass Index (BMI) < 30 kg/m² (according to medical record data)
* DLFT: diagnostic criteria for established or probable DLFT

Exclusion Criteria:

* Persons not affiliated with or not covered by a social security scheme
* Persons subject to legal protection measures (guardianship, trusteeship)
* Persons subject to judicial protection measures
* Pregnant women, women in labour or breastfeeding women
* MMSE score < 15 and/or MoCA score < 10
* Known COVID-19 infection within 6 months prior to inclusion
* Active smokers (> 4 cigarettes per day on a regular basis)
* Subject with a pacemaker (contraindication for bioelectrical impedance analysis)
* Subject with diabetes (type 1 or type 2)
* Taking medication (during the study) that interferes with taste

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Average latency of taste evoked potentials | After a fasting period of at least two hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France